CLINICAL TRIAL: NCT05492565
Title: A Study to Evaluate Clinical Benefits and Drawbacks of Antiretroviral Drugs as Pre-exposure Prophylaxis to Prevent HIV Infection Under Real-life Conditions Among Persons Who Pursue High-risk Sexual Practices: The Seville HIV PrEP Cohort
Brief Title: Seville Cohort of People at Substantial Risk for HIV Infection on Pre-exposure Prophylaxis
Acronym: SeVIHPrEP
Status: Enrolling by invitation | Type: Observational
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Collaborators: Instituto de Biomedicina de Sevilla (Unknown)
Responsible Party: Principal Investigator, Karin Neukam, Senior Investigator, Hospitales Universitarios Virgen del Rocío
Other Study IDs: SeVIHPrEP Cohort; FIS-PRE-2022-01 (Other: FISEVI)
Record Dates: First submitted 2022-07-30; First posted 2022-08-08 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: HIV Infection Primary; Hepatitis, Viral, Human; Sexually Transmitted Infections, Excluding HIV and Hepatitis
Keywords: PrEP; tenofovir disoproxyl fumarate; emtricitabine; HIV; Treponema pallidum; Neisseria gonorrhoeae; Chlamydia trachomatis; Mycoplasma genitalium; human papillomavirus; men who have sex with men; ChemSex
MeSH Terms: conditions — Hepatitis, Viral, Human; Sexually Transmitted Diseases; Hepatitis; Treponemal Infections; Homosexuality; Chemsex | interventions — Tenofovir; Tablets; Emtricitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — anal-rectal, oral and/or urethral exudate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Men who have sex with men: Men who have sex with men at substantial risk for HIV infection due to high-risk sexual habits
  Interventions: Drug: Tenofovir Disoproxil Fumarate 300 MG Oral Tablet
- Transgender women: Transgender women at substantial risk for HIV infection due to high-risk sexual habits
  Interventions: Drug: Tenofovir Disoproxil Fumarate 300 MG Oral Tablet
- Sex workers: Sex workers at substantial risk for HIV infection due to high-risk sexual habits
  Interventions: Drug: Tenofovir Disoproxil Fumarate 300 MG Oral Tablet
- HIV-uninfected people at substantial risk for HIV infection (other): All HIV-uninfected people at substantial risk for HIV infection due to any other reason, including having an HIV-positive life partnerwith an HIV-positive life partner
  Interventions: Drug: Tenofovir Disoproxil Fumarate 300 MG Oral Tablet

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate 300 MG Oral Tablet — Pre-exposure prophylaxis with coformulated Tenofovir Disoproxil Fumarate 300mg/Emtricitabine 200mg oral QD to prevent HIV infection
  Other Names: Emtricitabine 200 MG Oral Tablet

SUMMARY:
Pre-exposure prophylaxis (PrEP) based on tenofovir represents a considerably new preventive intervention that has shown to significantly decrease the number of HIV infections while it enables early diagnosis of HIV and other sexually transmitted diseases (STI).

In Southern Spain, the target population to receive PrEP are men who have sex with men (MSM) with a history of STI and who pursue high-risk sexual practices regarding the acquisition of HIV, including an elevate number of sex partners, no or inconsistent condom use and the use of specific recreational drugs in the context of sexual activity ("chemsex").

Despite the benefits of PrEP use, it must be taken into consideration that risk compensations that may facilitate the acquisition of other STI may occur, including a higher implementation of risk practices and an increase in the number of partners, which is made easy as various social networks designed for this purpose are available nowadays.

In order to better understand the benefit/drawback ratio, accurate data of a population using PrEP under real-life conditions, with densely scheduled follow-up and well-characterized (socio-)demographic parameters, sexual behaviour and STI are warranted.

DETAILED DESCRIPTION:
To date, the availability of highly-active antiretroviral drugs enables an efficient and persistent suppression of HIV replication. This, on the one hand, results in a considerably higher life expectancy and quality of life among persons living with HIV (PLWH) and, on the other hand, reduces the risk of viral transmission. Based on these advances, the Joint United Nations Programme on HIV/AIDS (UNAIDS) has developed strategies aiming to end the HIV/AIDS epidemic by including preventive tools. With the aim to prevent the acquisition of HIV infection, recommendations for the use of post-exposure prophylaxis were established, however, this strategy requires both the awareness of having been exposed to the virus, as well as the access to treatment within 72 hours after exposure, which represents important limitations when put into practice. To overcome these obstacles, pre-exposure prophylaxis has been implemented during the last decade.

PrEP represents a preventive intervention that has demonstrated a significant decrease in HIV infections in a large number of randomized clinical trials and observational studies among various populations. Apart from the preventive benefits, it furthermore supports the early diagnosis of HIV and other sexually transmitted diseases (STI), leading to the World Health Organisation (WHO) to recommend its use in 2012. As a result of a complex analysis including efficacy, risks and costs, PrEP was only recommended for persons at substantial risk to get infected. Main representatives are men who have sex with men (MSM), in whom a decrease of 44%-86% in HIV infection in pilot clinical trials was observed, as well as transgender women and persons with an HIV-positive partner. Among those compliant to daily PrEP, infection rates become close to zero. Although the majority of the guidelines are based on this modality, there is evidence that MSM showing less frequent sexual activity could also benefit from on-demand PrEP. In comparison with daily PrEP, the on-demand modality encourages adherence due to its contemporaneous use with the sexual intercourse.

So far, the WHO recommendations have been adapted in clinical guidelines of more than 60% of the countries worldwide, showing an increasing trend and promising results, as reported from ongoing PrEP programmes. In Spain, the use of PrEP based on tenofovir (TNF) and emtricitabine has demonstrated its benefit in a study to evaluate PrEP implementation in four Spanish settings. Subsequently, the Interministerial Commission for Medical Costs of the Spanish government approved financial support for PrEP in specific risk groups for HIV acquisition as defined by the National AIDS Plan (Plan Nacional sobre el SIDA, PNS) and since September of 2019, PrEP represents an integral part of the Andalusian Health System services. In this context, PrEP is offered as complementary preventive tool included in a package aimed to raise awareness in persons at high risk for HIV infection in order to break the chain of transmission and warrant required health care. Thus, in the setting of Seville, Andalusia (Spain), the main candidates to receive PrEP are MSM with a history of STI and high-risk sexual behaviour, including an elevated number of sex partners, no or rare use of condoms and chemsex. The latter refers to a relatively new trend in the MSM community and describes the use of specific recreational drugs, mainly metamphetamine, mephedrone, poppers or gammahydroxybutyrate (GHB)/gammabutyrolactone (GBL) in any combination or route of administration, in the context of sexual activity with one, but often multiple partners. Chemsex is associated with high-risk sex practices and the acquisition of STI.

Despite the high interest in this preventive tool, real-life data on PrEP use are scarce, the sexual habits among its users are not well characterised and there is no information available for Andalusia, and especially the region of Seville, where the number of candidates for PrEP is estimated to exceed 1000 according to the Andalusian Plan against HIV/AIDS and other STI (Plan Andaluz frente al VIH/SIDA y otras ITS, PASIDA). Likewise, while the of primary HIV infections during PrEP are likely rare-to-absent, they cannot be excluded and their characteristics and clinical management are poorly studied. Additionally, in spite of the benefit of PrEP, there are various considerations regarding its use, like the development of adverse events on the short or long term in healthy people taking antiretroviral drugs, as in the case of TNF, renal function and bone density may be affected. Another major concern is the possibility of risk compensation in persons who feel less vulnerable due to the protective effect of PrEP. This could be manifested in a shift of sexual habits towards high-risk behaviour and/or an increase in the number of sex partners which can be achieved comfortably while remaining anonymous, given the social networks designed for this purpose available nowadays. Consequently, transmission of other STI, unintended pregnancies and resistance to TNF in case of primary HIV infection would be encouraged. Studies under real-life conditions including frequent and detailed monitoring are strongly needed in order to gain knowledge on the possible impact of PrEP on its users, taking into account possible changes in life style caused by the constant evolution of society and social media, like dating applications. In fact, a change in the social profile of MSM newly diagnosed with HIV infection has been reported recently in Madrid, which supports the need to improve the characterization and motorization of those participating in PrEP programmes.

In order to clarify this issue, accurate data of a population using PrEP under real-life conditions, with densely scheduled follow-up and well-characterized (socio-)demographic parameters, sexual behaviour and STI are warranted.

ELIGIBILITY:
Inclusion Criteria:

* HIV negative as demonstrated by negative HIV serology as determined by EIA and Western-Blot.
* Older than 18 years.
* At high risk of acquiring HIV infection by sexual transmission.
* MSM and transsexual persons who met at least two of the following criteria during the year prior to visit:
* More than ten different sexual partners.
* Anal sexual intercourse without using a condom.
* Consumption of drugs in order to establish and/or maintain sexual relations without condom.
* Administration of post-exposition prophylaxis in various occasions de profilaxis post- exposición en varias ocasiones.
* At least one bacterial STI.
* Women who prostitute themselves with no or irregular use of a condom. -Start daily or on-demand PrEP with TDF/FTC.
* Give their written informed consent to participate in the cohort and its substudies.

Exclusion Criteria:

* Glomerular filtration rate <60 ml/min.
* For on-demand PrEP: diagnosis of chronic hepatitis B.
* Allergic to TDF and/or FTC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants of the SeVIHPrEP cohort are recruited from the candidates for a PrEP programme derived from the outpatient STI clinic at the Clinical Unit of Infecious Diseases and Preventive Medicine (Unidad Clínica de Enfermedades Infecciosas y Medicina Preventiva, UCEIMP) of the Virgen del Rocío University Hospital (Hospital Universitario Virgen del Rocío) in Seville, Spain. Candidates are informed about the SeVIHPrEP protocol, an information sheet is handed out and additionally, the study is explained by the physician. They are then invited to participate in the cohort and upon acceptance, are asked to sign a written informed consent.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline proportion of PrEP users with STI-4c at one year | Baseline through one year
  Analysis of a change in the proportion of persons that present with infection by at least one of the following four common sexually transmitted pathogens (STI-4c): Treponema pallidum, Neisseria gonorrhoeae, Chlamydia trachomatis and/or Mycoplasma genitalium.
Incidence of primary HIV infection | Through study completion (an average 3 years)
  Determination of the incidence of primary HIV infections during PrEP use

SECONDARY OUTCOMES:
Proportion of PrEP users with STI other than STI-4c or HIV | Through study completion (an average 3 years)
  Determination of the proportion of persons that present with STI other than those analysed in the primary outcome
Number of STI | Through study completion (an average 3 years)
  Determination of the number of STI PrEP users present with STI at the scheduled visits
Incidences of STI other than HIV | Through study completion (an average 3 years)
  Determination of the incidences of individual STI other than HIV
Sexual behaviour | Through study completion (an average 3 years)
  Determination of the number of distinct sexual risk practices conducted per person since the last study visit
Adverse events | Through study completion (an average 3 years)
  Determination of the rate of adverse events related to the antiretroviral drugs used for PrEP
Adherence to PrEP | Through study completion (an average 3 years)
  Evaluation of the adherence to PrEP modalities (daily PrEP: proportion of days PrEP was taken; on-demand PrEP: proportion of sexual intercourse with PrEP)
Predictors of the incidence of HIV and other STI | Through study completion (an average 3 years)
  Identification of factors associated with the incidence of HIV infection and STI other than HIV
Predictors of a change in the proportion of STI-4c | Baseline through one year
  Identification of factors associated with a change in the proportion of STI-4c

CONTACTS AND LOCATIONS:
Overall Officials: Karin Neukam, PharmD, PhD, Study Director — Instituto de Biomedicina de Sevilla/ H Universitario Virgen del Rocío/ CSIC/ Universidad de Sevilla; César Sotomayor de la Piedra, MD, Principal Investigator — Hospitales Universitarios Virgen del Rocío; Marta Herrero Romero, MD, PhD, Principal Investigator — Hospitales Universitarios Virgen del Rocío; Alicia Gutiérrez Valencia, PharmD, PhD, Principal Investigator — Instituto de Biomedicina de Sevilla/ H Universitario Virgen del Rocío/ CSIC/ Universidad de Sevilla; Luis F López-Cortés, MD, PhD, Principal Investigator — Instituto de Biomedicina de Sevilla/ H Universitario Virgen del Rocío/ CSIC/ Universidad de Sevilla
Locations (1):
- Virgen del Rocío University Hospital, Seville, Andalusia, Spain

REFERENCES:
- [Background] Donnell D, Baeten JM, Kiarie J, Thomas KK, Stevens W, Cohen CR, McIntyre J, Lingappa JR, Celum C; Partners in Prevention HSV/HIV Transmission Study Team. Heterosexual HIV-1 transmission after initiation of antiretroviral therapy: a prospective cohort analysis. Lancet. 2010 Jun 12;375(9731):2092-8. doi: 10.1016/S0140-6736(10)60705-2. Epub 2010 May 26. PMID 20537376
- [Background] Cohen MS, Chen YQ, McCauley M, Gamble T, Hosseinipour MC, Kumarasamy N, Hakim JG, Kumwenda J, Grinsztejn B, Pilotto JH, Godbole SV, Chariyalertsak S, Santos BR, Mayer KH, Hoffman IF, Eshleman SH, Piwowar-Manning E, Cottle L, Zhang XC, Makhema J, Mills LA, Panchia R, Faesen S, Eron J, Gallant J, Havlir D, Swindells S, Elharrar V, Burns D, Taha TE, Nielsen-Saines K, Celentano DD, Essex M, Hudelson SE, Redd AD, Fleming TR; HPTN 052 Study Team. Antiretroviral Therapy for the Prevention of HIV-1 Transmission. N Engl J Med. 2016 Sep 1;375(9):830-9. doi: 10.1056/NEJMoa1600693. Epub 2016 Jul 18. PMID 27424812
- [Background] Smith DK, Grohskopf LA, Black RJ, Auerbach JD, Veronese F, Struble KA, Cheever L, Johnson M, Paxton LA, Onorato IM, Greenberg AE; U.S. Department of Health and Human Services. Antiretroviral postexposure prophylaxis after sexual, injection-drug use, or other nonoccupational exposure to HIV in the United States: recommendations from the U.S. Department of Health and Human Services. MMWR Recomm Rep. 2005 Jan 21;54(RR-2):1-20. PMID 15660015
- [Background] Guideline on When to Start Antiretroviral Therapy and on Pre-Exposure Prophylaxis for HIV. Geneva: World Health Organization; 2015 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK327115/ PMID 26598776
- [Background] Molina JM, Capitant C, Spire B, Pialoux G, Cotte L, Charreau I, Tremblay C, Le Gall JM, Cua E, Pasquet A, Raffi F, Pintado C, Chidiac C, Chas J, Charbonneau P, Delaugerre C, Suzan-Monti M, Loze B, Fonsart J, Peytavin G, Cheret A, Timsit J, Girard G, Lorente N, Preau M, Rooney JF, Wainberg MA, Thompson D, Rozenbaum W, Dore V, Marchand L, Simon MC, Etien N, Aboulker JP, Meyer L, Delfraissy JF; ANRS IPERGAY Study Group. On-Demand Preexposure Prophylaxis in Men at High Risk for HIV-1 Infection. N Engl J Med. 2015 Dec 3;373(23):2237-46. doi: 10.1056/NEJMoa1506273. Epub 2015 Dec 1. PMID 26624850
- [Background] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279
- [Background] Spinner CD, Boesecke C, Zink A, Jessen H, Stellbrink HJ, Rockstroh JK, Esser S. HIV pre-exposure prophylaxis (PrEP): a review of current knowledge of oral systemic HIV PrEP in humans. Infection. 2016 Apr;44(2):151-8. doi: 10.1007/s15010-015-0850-2. Epub 2015 Oct 15. PMID 26471511
- [Background] Antoni G, Tremblay C, Delaugerre C, Charreau I, Cua E, Rojas Castro D, Raffi F, Chas J, Huleux T, Spire B, Capitant C, Cotte L, Meyer L, Molina JM; ANRS IPERGAY study group. On-demand pre-exposure prophylaxis with tenofovir disoproxil fumarate plus emtricitabine among men who have sex with men with less frequent sexual intercourse: a post-hoc analysis of the ANRS IPERGAY trial. Lancet HIV. 2020 Feb;7(2):e113-e120. doi: 10.1016/S2352-3018(19)30341-8. Epub 2019 Nov 26. PMID 31784343
- [Background] Schaefer R, Schmidt HA, Ravasi G, Mozalevskis A, Rewari BB, Lule F, Yeboue K, Brink A, Mangadan Konath N, Sharma M, Seguy N, Hermez J, Alaama AS, Ishikawa N, Dongmo Nguimfack B, Low-Beer D, Baggaley R, Dalal S. Adoption of guidelines on and use of oral pre-exposure prophylaxis: a global summary and forecasting study. Lancet HIV. 2021 Aug;8(8):e502-e510. doi: 10.1016/S2352-3018(21)00127-2. Epub 2021 Jul 12. PMID 34265283
- [Background] Reitsema M, Hoek AJV, van der Loeff MS, Hoornenborg E, van Sighem A, Wallinga J, van Benthem B, Xiridou M. Preexposure prophylaxis for men who have sex with men in the Netherlands: impact on HIV and Neisseria gonorrhoeae transmission and cost-effectiveness. AIDS. 2020 Mar 15;34(4):621-630. doi: 10.1097/QAD.0000000000002469. PMID 31895142
- [Background] Iniesta C, Coll P, Barbera MJ, Garcia Deltoro M, Camino X, Fagundez G, Diaz A, Polo R; Spanish Working Group for PrEP. Implementation of pre-exposure prophylaxis programme in Spain. Feasibility of four different delivery models. PLoS One. 2021 Feb 8;16(2):e0246129. doi: 10.1371/journal.pone.0246129. eCollection 2021. PMID 33556085
- [Background] Maxwell S, Shahmanesh M, Gafos M. Chemsex behaviours among men who have sex with men: A systematic review of the literature. Int J Drug Policy. 2019 Jan;63:74-89. doi: 10.1016/j.drugpo.2018.11.014. Epub 2018 Dec 1. PMID 30513473
- [Background] Guerras JM, Hoyos Miller J, Agusti C, Chanos S, Pichon F, Kuske M, Cigan B, Fuertes R, Stefanescu R, Ooms L, Casabona J, de la Fuente L, Belza MJ; Euro HIV EDAT Working Group. Association of Sexualized Drug Use Patterns with HIV/STI Transmission Risk in an Internet Sample of Men Who Have Sex with Men from Seven European Countries. Arch Sex Behav. 2021 Feb;50(2):461-477. doi: 10.1007/s10508-020-01801-z. Epub 2020 Sep 2. PMID 32875382
- [Background] Ambrosioni J, Petit E, Liegeon G, Laguno M, Miro JM. Primary HIV-1 infection in users of pre-exposure prophylaxis. Lancet HIV. 2021 Mar;8(3):e166-e174. doi: 10.1016/S2352-3018(20)30271-X. Epub 2020 Dec 11. PMID 33316212
- [Background] Adams JL, Shelley K, Nicol MR. Review of Real-World Implementation Data on Emtricitabine-Tenofovir Disoproxil Fumarate as HIV Pre-exposure Prophylaxis in the United States. Pharmacotherapy. 2019 Apr;39(4):486-500. doi: 10.1002/phar.2240. Epub 2019 Apr 1. PMID 30815960
- [Background] Barreiro P. Sexually Transmitted Infections on the Rise in PrEP Users. AIDS Rev. 2018 Jan-Mar;20(1):71. PMID 29628512
- [Background] Ayerdi Aguirrebengoa O, Vera Garcia M, Arias Ramirez D, Gil Garcia N, Puerta Lopez T, Clavo Escribano P, Ballesteros Martin J, Lejarraga Canas C, Fernandez Pineiro N, Fuentes Ferrer ME, Garcia Lotero M, Hurtado Gallegos E, Raposo Utrilla M, Estrada Perez V, Del Romero Guerrero J, Rodriguez Martin C. Low use of condom and high STI incidence among men who have sex with men in PrEP programs. PLoS One. 2021 Feb 4;16(2):e0245925. doi: 10.1371/journal.pone.0245925. eCollection 2021. PMID 33539363
- [Background] Di Ciaccio M, Sagaon-Teyssier L, Mimi M, Suzan-Monti M, Protiere C, Rojas Castro D, Meyer L, Tremblay C, Chidiac C, Capitant C, Preau M, Molina JM, Spire B; ANRS IPERGAY Study Group. Changes in Sexual Behaviors in Men Who Have Sex with Men: A Comparison Between the Double-Blind and Open-Label Extension Phases of the ANRS-IPERGAY Trial. AIDS Behav. 2020 Nov;24(11):3093-3106. doi: 10.1007/s10461-020-02864-8. PMID 32306213
- [Background] Ayerdi Aguirrebengoa O, Vera Garcia M, Puerta Lopez T, Clavo Escribano P, Ballesteros Martin J, Lejarrag Canas C, Fuentes Ferrer E, Raposo Utrilla M, Estrada Perez V, Del Romero Guerrero J, Rodriguez Martin C; Sandoval Study Group. Changes in the profile of newly HIV-diagnosed men who have sex with men, Madrid, 2014 to 2019. Euro Surveill. 2021 Nov;26(47):2001501. doi: 10.2807/1560-7917.ES.2021.26.47.2001501. PMID 34823642
- See also: United Nations Programme on HIV/AIDS 2020. 90-90-90: An ambitious treatment target to help end the AIDS epidemic. 2019 — https://www.unaids.org/sites/default/files/media_asset/90-90-90_en.pdf
- See also: Ministerio de Sanidad Servicios Sociales e Igualdad. Documento de consenso. Profilaxis Preexposición al VIH en España. Plan Nacional sobre el Sida. Published Online First: 2018 — http://www.mscbs.gob.es/ciudadanos/enfLesiones/enfTransmisibles/sida/docs/PROFILAXIS_PREEXPOSICION_VIH.pdf